# **BPIT\_2024\_ICF: Informed Consent Form**

**Study Title:** A Prospective, Single-Center, Interventional Study to Evaluate the 5-Line Principle of Balanced Intensity Training (BPIT) for Enhancing Physical Performance and Reducing Injury Risk

Protocol ID: BPIT-GFFI-2024-001

**Principal Investigator:** Dr. Neeraj Mehta, PhD **Contact:** [6148228038] / [Info@mmsxauthority.com]

Document Created Date: 07 May, 2024

Site: GFFI Fitness Academy, [35, NWA, Punjabi Bagh, West, New Delhi 110026]

## What is the purpose of the study?

This is a 6-week training study to test a new exercise method called Balanced Progression Intensity Training (BPIT) based on the 5-Line Principle. We want to see if it improves strength and reduces injury risk compared to your current fitness level.

## Who is doing the study?

The study is sponsored by MMSx Authority Institute for Movement Mechanics & Biomechanics Research Inc. and conducted at GFFI Fitness Academy under the direction of Dr. Neeraj Mehta.

## What will happen if I take part?

- You will train 3 times per week (60-minute sessions) for 6 weeks (total 18 sessions).
- Each session follows the BPIT 5-Line progression (ground-based → knee-level → standing → head-level → plyometric).
- Before starting and after Week 6 we will measure: Your maximum strength (1RM squat, bench press, deadlift) Heart rate and heart rate variability Muscle activation with surface EMG Knee and spine angles with video analysis
- You will be asked to report any discomfort or injury immediately.

## How many people will take part?

23 healthy adults.

## What are the risks and discomforts?

Possible muscle soreness, fatigue, or minor strains (risk similar to normal gym training). Serious injury is very rare. A qualified trainer will supervise every session. You can stop at any time.

#### Are there benefits?

You will receive 6 weeks of free supervised training and detailed personal fitness assessment (worth several thousand rupees).

# Will my information be kept confidential?

Yes. Your name will be replaced by a code. Only the study team will have access to the link between code and name. Results will be published/presented only in summary form.

# Can I leave the study?

Yes, at any time without giving a reason and without any consequence.

# **Costs and compensation**

No cost to you. You will receive [state any compensation or "no financial compensation – only free training and testing"].

# Who do I contact if I have questions?

Dr. Neeraj Mehta – **Contact:** [6148228038] / [Info@mmsxauthority.com]

In case of injury: same contact or visit nearest medical facility (costs covered by sponsor if directly related to study).

## **Participant Statement**

| I have read this form, had the ch | ance to ask questions, and volunt | arily agree to take part. |
|---|---|---|
| Name: | Signature: | Date: |
| If participant <18 years: Parent/0 | Guardian signature | |
| Investigator Statement | | |
| I have explained the study and a | answered all questions. | |
| Signature Dr. Neeraj Mehta | Date | |